CLINICAL TRIAL: NCT01319565
Title: A Prospective Randomized Study of Cell Transfer Therapy for Metastatic Melanoma Using Short-Term Cultured Tumor-Infiltrating Lymphocytes Plus IL-2 Following Either a Non-Myeloablative Lymphocyte Depleting Chemotherapy Regimen Alone or in Conjunction With 12Gy Total Body Irradiation (TBI)
Brief Title: Prospective Randomized Study of Cell Transfer Therapy for Metastatic Melanoma Using Tumor Infiltrating Lymphocytes Plus IL-2 Following Non-Myeloablative Lymphocyte Depleting Chemo Regimen Alone or in Conjunction With 12Gy Total Body Irradiation (TBI...
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: National Cancer Institute (NCI) (NIH)
Responsible Party: Principal Investigator, Steven Rosenberg, M.D., Principal Investigator, National Cancer Institute (NCI)
Organization: National Institutes of Health Clinical Center (CC) (NIH)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 110123; 11-C-0123
Record Dates: First submitted 2011-03-18; First posted 2011-03-21 (Estimated); Results first posted 2025-12-19 (Actual); Last update posted 2025-12-19 (Actual); Status verified 2025-12

CONDITIONS: Metastatic Melanoma; Skin Cancer
Keywords: Young TIL; Metastatic Melanoma; Immunotherapy; Adoptive Cell Therapy; Skin Cancer
MeSH Terms: conditions — Melanoma; Skin Neoplasms | interventions — aldesleukin; Interleukin-2; Cyclophosphamide; fludarabine; fludarabine phosphate; Whole-Body Irradiation

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Arm 1/Adoptive Cell Therapy (ACT) (Experimental): Non-myeloablative lymphodepleting preparative regimen of cyclophosphamide and fludarabine + young tumor infiltrating lymphocytes (TIL) + high dose aldesleukin
  Interventions: Drug: Aldesleukin; Drug: Cyclophosphamide; Drug: Fludarabine; Biological: Young TIL
- Arm 2/Adoptive Cell Therapy (ACT) + Total Body Irradiation (TBI) (Experimental): Non-myeloablative lymphodepleting preparative regimen of cyclophosphamide and fludarabine + young tumor infiltrating lymphocytes (TIL) + high dose aldesleukin + total body irradiation (TBI)
  Interventions: Drug: Aldesleukin; Drug: Cyclophosphamide; Drug: Fludarabine; Biological: Young TIL; Radiation: Total Body Irradiation (TBI)

INTERVENTIONS:
Drug: Aldesleukin — Arm 1 and Arm 2 - Days 1 to 4: Aldesleukin 720,000 IU/kg intravenous (IV) (based on total body weight) over 15 minutes every eight hours (+/- 1 hour) for up to 5 days (maximum 15 doses).
  Other Names: Interleukin-2
Drug: Cyclophosphamide — Arm 1 and Arm 2 - Days -7 and -6: Cyclophosphamide 60 mg/kg/day X 2 days intravenous (IV) in 250 mL dextrose 5% in water (D5W) with Mesna 15 mg/kg/day X 2 days over 1 hr.
  Other Names: Cytoxan
Drug: Fludarabine — Arm 1 and Arm 2 - Days -7 to -3: Fludarabine 25 mg/m^2/day intravenous piggyback (IVPB) daily over 15-30 minutes for 5 days.
  Other Names: Fludara
Biological: Young TIL — Arm 1 and Arm 2 - Day 0: Cells will be infused intravenously (IV) on the Patient Care Unit over 20-30 minutes.
  Other Names: Young tumor infiltrating lymphocytes
Radiation: Total Body Irradiation (TBI) — Arm 2 - Days -3 to -1: Ondansetron 0.15 mg/kg intravenous (IV) x 1 dose pre-total body irradiation (TBI). Patients will then receive 2 Gray (Gy) TBI twice a day for 3 days (total dose 12 Gy using a linear accelerator in Radiation Oncology.
  Other Names: TBI
  Arms: Arm 2/Adoptive Cell Therapy (ACT) + Total Body Irradiation (TBI)

SUMMARY:
Background:

- An experimental treatment for metastatic melanoma involves cell therapy, in which researchers take white blood cells (lymphocytes) from the tumor tissue, grow them in the laboratory in large numbers, and then use the cells to attack the tumor tissue. Before receiving the cells, chemotherapy is needed to temporarily suppress the immune system to improve the chances that the tumor-fighting cells will be able to survive in the body. In some studies of cell therapy, individuals who have received total body irradiation (TBI) in addition to the chemotherapy (in order to increase the length of time that they do not produce white blood cells) seem to have a slightly better response to the treatment, but it is not known if adding radiation to the cell therapy will cause a better response for all individuals. Researchers are interested in comparing cell therapy given with the usual chemotherapy to cell therapy given with the usual chemotherapy and TBI.

Objectives:

- To compare the effectiveness of cell therapy given with chemotherapy to cell therapy given with chemotherapy and total body irradiation in individuals with metastatic melanoma.

Eligibility:

- Individuals at least 18 years of age who have been diagnosed with metastatic melanoma.

Design:

* Participants will be screened with a physical examination, medical history, blood tests, and tumor imaging studies.
* Participants will be divided into two groups: cell therapy with chemotherapy alone (group 1) or cell therapy with chemotherapy plus TBI (group 2).
* All participants will provide a tumor sample from either surgery or a tumor biopsy for white blood cell collection.
* Participants will have leukapheresis to collect additional white blood cells for cell growth and future testing, and TBI group participants will also provide stem cells to help them recover after radiation. (TBI participants who cannot provide enough stem cells will be moved to the non-radiation treatment group.)
* Participants will have chemotherapy with cyclophosphamide (two treatments over 2 days) and fludarabine (five treatments over 5 days) starting 7 days before the cell therapy. Participants in the TBI group will also have TBI for the 3 days immediately before the cell therapy.
* All participants will receive the white blood cells, followed by high dose aldesleukin every 8 hours for up to 5 days after the cell infusion to help keep the therapy cells alive and active. Participants will also have injections of filgrastim to stimulate blood cell production, and participants in the TBI group will also receive their stem cells.
* Participants will take an antibiotic for at least 6 months after treatment to prevent pneumonia and will be asked to return for regular monitoring and follow-up visits for at least 5 years to evaluate the tumors response to treatment.

DETAILED DESCRIPTION:
Background:

* Adoptive cell therapy (ACT) using autologous tumor infiltrating lymphocytes can mediate the regression of bulky metastatic melanoma when administered along with high-dose aldesleukin (IL-2) following a non-myeloablative lymphodepleting chemotherapy preparative regimen consisting of cyclophosphamide and fludarabine.
* In a series of consecutive trials using this chemotherapy preparative regimen alone or with 2 Gray (Gy) or 12 Gy total body irradiation (TBI) objective response rates using Response Evaluation Criteria in Solid Tumors (RECIST) criteria were 49%, 52%, and 72%, respectively. Complete regression rates in these three consecutive trials were 12%, 20%, and 40%, respectively strongly suggesting that the addition of TBI could improve the complete regression rate. Of the 20 complete regressions seen in this trial, 19 are on-going at 37 to 82 months.
* Because of the complexity of developing selected TIL for use in adoptive transfer, we have recently developed a simplified method for producing TIL that is more applicable to use in outside institutions. Utilizing young TIL cells (sometimes with cluster of differentiation 8 (CD8) purification) in 105 patients, the objective response rate was 34% with a 6.6 % incidence of complete regressions. All patients in this trial received the cyclophosphamide fludarabine regimen alone.
* Because of the strong suggestion that the addition of TBI to the chemotherapy regimen could increase durable, complete regression rates in patients with metastatic melanoma, we are now attempting to definitively determine whether the addition of TBI to the chemotherapy preparative regimen can improve complete response rates, and overall survival in patients receiving young TIL.

Objectives:

-To determine, in a prospective randomized trial, the complete response rate and survival of patients with metastatic melanoma receiving adoptive cell transfer (ACT) using young TIL plus aldesleukin treatment following either a chemotherapy preparative regimen alone, or the same chemotherapy preparative regimen plus TBI.

Eligibility:

-Patients who are 18 years or older must have:

* Evaluable metastatic melanoma;
* Metastatic melanoma lesion suitable for surgical resection for the preparation of TIL;
* No contraindications to high dose aldesleukin administration or total body irradiation;
* No concurrent major medical illnesses or any form of immunodeficiency

Design:

-Patients with metastatic melanoma will have lesions resected and after TIL growth is established patients with will be prospectively randomized to receive ACT with young TIL plus aldesleukin following either a non-myeloablative chemotherapy preparative regimen or this same regimen plus TBI.

ELIGIBILITY:
* INCLUSION CRITERIA:

  1. Measurable metastatic melanoma with at least one lesion that is resectable for tumor infiltrating lymphocytes (TIL) generation. The lesion must be of at least 1cm in diameter that can be surgically removed with minimal morbidity (defined as any operation for which expected hospitalization less than or equal to 7 days).
  2. Patients with 3 or less brain metastases are eligible. Note: If lesions are symptomatic or greater than or equal to 1 cm each, these lesions must have been treated and stable for 3 months for the patient to be eligible.
  3. Greater than or equal to 18 years of age and less than or equal to 66 years of age.
  4. Willing to practice birth control during treatment and for four months after receiving all protocol related therapy.
  5. Life expectancy of greater than three months
  6. Willing to sign a durable power of attorney.
  7. Able to understand and sign the Informed Consent Document
  8. Clinical performance status of eastern Cooperative Oncology Group (ECOG) 0 or 1.
  9. Hematology:
* Absolute neutrophil count greater than 1000/mm(3)
* Hemoglobin greater than 8.0 g/dl
* Platelet count greater than 100,000/mm(3)

  j. Serology:
* Seronegative for human immunodeficiency virus (HIV) antibody. (The experimental treatment being evaluated in this protocol depends on an intact immune system. Patients who are HIV seropositive can have decreased immune competence and thus be less responsive to the experimental treatment and more susceptible to its toxicities.)
* Seronegative for hepatitis B antigen, or hepatitis C antibody or antigen.

  k. Chemistry:
* Serum alanine aminotransferase (ALT)/aspartate aminotransferase (AST) less than three times the upper limit of normal.
* Calculated creatinine clearance (eGFR) > 50 ml/min.
* Total bilirubin less than or equal to 2 mg/dl, except in patients with

Gilbert's Syndrome who must have a total bilirubin less than 3 mg/dl.

l. More than four weeks must have elapsed since any prior systemic therapy at the time of randomization, and patient's toxicities must have recovered to a grade 1 or less (except for alopecia or vitiligo). Patients must have stable or progressing disease after prior treatment.

Note: Patients may have undergone minor surgical procedures within the past 3 weeks, as long as all toxicities have recovered to grade 1 or less or as specified in the inclusion criteria.

m. Six weeks must have elapsed since any prior anti-cytotoxic T-lymphocyte associated protein 4 (CTLA4) antibody therapy to allow antibody levels to decline.

Note: Patients who have previously received ipilimumab or tremelimumab, anti-programmed cell death protein 1 (PD1) or anti-programmed cell death ligand 1 (PD-L1) antibodies and have documented gastrointestinal (GI) toxicity must have a normal colonoscopy with normal colonic biopsies.

EXCLUSION CRITERIA:

1. Prior cell transfer therapy which included a non-myeloablative or myeloablative chemotherapy regimen.
2. Women of child-bearing potential who are pregnant or breastfeeding because 10 of the potentially dangerous effects of the preparative chemotherapy on the fetus or infant.
3. Systemic steroid therapy requirement.
4. Active systemic infections, coagulation disorders or other active major medical illnesses of the cardiovascular, respiratory or immune system, as evidenced by a positive stress thallium or comparable test, myocardial infarction, cardiac arrhythmias, obstructive or restrictive pulmonary disease.
5. Any form of primary immunodeficiency (such as Severe Combined Immunodeficiency Disease and acquired immunodeficiency syndrome (AIDS).
6. Opportunistic infections (The experimental treatment being evaluated in this protocol depends on an intact immune system. Patients who have decreased immune competence may be less responsive to the experimental treatment and more susceptible to its toxicities.)
7. History of severe immediate hypersensitivity reaction to any of the agents used in this study.
8. History of coronary revascularization or ischemic symptoms.
9. Any patient known to have a left ventricular ejection fraction (LVEF) less than or equal to 45%.
10. In patients > 60 years old, documented LVEF of less than or equal to 45%.
11. Documented forced expiratory volume in one second (FEV1) less than or equal to 60% predicted tested in patients with:

    * A prolonged history of cigarette smoking (20 pk/year of smoking within the past 2 years)
    * Symptoms of respiratory dysfunction
12. Prior radiation therapy that, in the judgment of the radiation oncologist, precludes the administration of total body irradiation.

Ages: 18 Years to 66 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 102 (Actual)
Dates: Start 2011-03-24 (Actual); Primary Completion 2024-09-10 (Actual); Study Completion 2024-09-10 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Steven A Rosenberg, M.D., Principal Investigator — National Cancer Institute (NCI)
Locations (1):
- National Institutes of Health Clinical Center, Bethesda, Maryland, United States

IPD SHARING:
Plan to Share IPD: Yes
All individual participant data (IPD) recorded in the medical record will be shared with intramural investigators upon request.
Supporting Information: Study Protocol, SAP, ICF
Time Frame: Clinical data available during the study and indefinitely.
Access Criteria: Clinical data will be made available via subscription to Biomedical Translational Research Information System (BTRIS) and with the permission of the study principal investigator (PI).

REFERENCES:
- [Background] Dudley ME, Yang JC, Sherry R, Hughes MS, Royal R, Kammula U, Robbins PF, Huang J, Citrin DE, Leitman SF, Wunderlich J, Restifo NP, Thomasian A, Downey SG, Smith FO, Klapper J, Morton K, Laurencot C, White DE, Rosenberg SA. Adoptive cell therapy for patients with metastatic melanoma: evaluation of intensive myeloablative chemoradiation preparative regimens. J Clin Oncol. 2008 Nov 10;26(32):5233-9. doi: 10.1200/JCO.2008.16.5449. Epub 2008 Sep 22. PMID 18809613
- [Background] Atkins MB, Lotze MT, Dutcher JP, Fisher RI, Weiss G, Margolin K, Abrams J, Sznol M, Parkinson D, Hawkins M, Paradise C, Kunkel L, Rosenberg SA. High-dose recombinant interleukin 2 therapy for patients with metastatic melanoma: analysis of 270 patients treated between 1985 and 1993. J Clin Oncol. 1999 Jul;17(7):2105-16. doi: 10.1200/JCO.1999.17.7.2105. PMID 10561265
- [Background] Rosenberg SA, Yannelli JR, Yang JC, Topalian SL, Schwartzentruber DJ, Weber JS, Parkinson DR, Seipp CA, Einhorn JH, White DE. Treatment of patients with metastatic melanoma with autologous tumor-infiltrating lymphocytes and interleukin 2. J Natl Cancer Inst. 1994 Aug 3;86(15):1159-66. doi: 10.1093/jnci/86.15.1159. PMID 8028037
- [Background] Goff SL, Dudley ME, Citrin DE, Somerville RP, Wunderlich JR, Danforth DN, Zlott DA, Yang JC, Sherry RM, Kammula US, Klebanoff CA, Hughes MS, Restifo NP, Langhan MM, Shelton TE, Lu L, Kwong ML, Ilyas S, Klemen ND, Payabyab EC, Morton KE, Toomey MA, Steinberg SM, White DE, Rosenberg SA. Randomized, Prospective Evaluation Comparing Intensity of Lymphodepletion Before Adoptive Transfer of Tumor-Infiltrating Lymphocytes for Patients With Metastatic Melanoma. J Clin Oncol. 2016 Jul 10;34(20):2389-97. doi: 10.1200/JCO.2016.66.7220. Epub 2016 May 23. PMID 27217459
- [Background] Seitter SJ, Sherry RM, Yang JC, Robbins PF, Shindorf ML, Copeland AR, McGowan CT, Epstein M, Shelton TE, Langhan MM, Franco Z, Danforth DN, White DE, Rosenberg SA, Goff SL. Impact of Prior Treatment on the Efficacy of Adoptive Transfer of Tumor-Infiltrating Lymphocytes in Patients with Metastatic Melanoma. Clin Cancer Res. 2021 Oct 1;27(19):5289-5298. doi: 10.1158/1078-0432.CCR-21-1171. PMID 34413159
- [Derived] Crompton JG, Sukumar M, Roychoudhuri R, Clever D, Gros A, Eil RL, Tran E, Hanada K, Yu Z, Palmer DC, Kerkar SP, Michalek RD, Upham T, Leonardi A, Acquavella N, Wang E, Marincola FM, Gattinoni L, Muranski P, Sundrud MS, Klebanoff CA, Rosenberg SA, Fearon DT, Restifo NP. Akt inhibition enhances expansion of potent tumor-specific lymphocytes with memory cell characteristics. Cancer Res. 2015 Jan 15;75(2):296-305. doi: 10.1158/0008-5472.CAN-14-2277. Epub 2014 Nov 28. PMID 25432172
- See also: NIH Clinical Center Detailed Web Page — https://clinicalstudies.info.nih.gov/cgi/detail.cgi?B_2011-C-0123.html

RESULTS

PARTICIPANT FLOW:
Groups:
- Arm 1: Tumor Infiltrating Lymphocytes (TIL) + High Dose (HD) Interleukin-2 (IL-2): Non-myeloablative lymphodepleting preparative regimen of cyclophosphamide and fludarabine + young tumor infiltrating lymphocytes (TIL) + high dose aldesleukin
  Aldesleukin: Arm 1 - Days 1 to 4: Aldesleukin 720,000 IU/kg intravenous (IV) (based on total body weight) over 15 minutes every eight hours (+/- 1 hour) for up to 5 days (maximum 15 doses).
  Cyclophosphamide: Arm 1 - Days -7 and -6: Cyclophosphamide 60 mg/kg/day X 2 days intravenous (IV) in 250 mL dextrose 5% in water (D5W) with Mesna 15 mg/kg/day X 2 days over 1 hr.
  Fludarabine: Arm 1 - Days -7 to -3: Fludarabine 25 mg/m^2/day intravenous piggyback (IVPB) daily over 15-30 minutes for 5 days.
  Young TIL: Arm 1 - Day 0: Cells will be infused intravenously (IV) on the Patient Care Unit over 20-30 minutes.
- Arm 2: Tumor Infiltrating Lymphocytes + High Dose Interleukin-2 + 1200 Total Body Irradiation (TBI): Non-myeloablative lymphodepleting preparative regimen of cyclophosphamide and fludarabine + young tumor infiltrating lymphocytes (TIL) + high dose aldesleukin + total body irradiation (TBI)
  Aldesleukin: Arm 2 - Days 1 to 4: Aldesleukin 720,000 IU/kg intravenous (IV) (based on total body weight) over 15 minutes every eight hours (+/- 1 hour) for up to 5 days (maximum 15 doses).
  Cyclophosphamide: Arm 2 - Days -7 and -6: Cyclophosphamide 60 mg/kg/day X 2 days intravenous (IV) in 250 mL dextrose 5% in water (D5W) with Mesna 15 mg/kg/day X 2 days over 1 hr.
  Fludarabine: Arm 2 - Days -7 to -3: Fludarabine 25 mg/m^2/day intravenous piggyback (IVPB) daily over 15-30 minutes for 5 days.
  Young TIL: Arm 2 - Day 0: Cells will be infused intravenously (IV) on the Patient Care Unit over 20-30 minutes.
  Total Body Irradiation (TBI): Arm 2 - Days -3 to -1: Ondansetron 0.15 mg/kg intravenous (IV) x 1 dose pre-total body irradiation (TBI). Patients will then receive 2 Gray (Gy) TBI twice a day for 3 days (total dose 12 Gy using a linear accelerator in Radiation Oncology.
- Arm 1X: Tumor Infiltrating Lymphocytes (TIL) + High Dose (HD) Interleukin-2 (IL-2): Arm 1X: Compassionate Exemption. Participant received young tumor infiltrating lymphocytes (TIL) and Interleukin-2 (IL-2), but not cyclophosphamide or fludarabine (they were administered before the participant enrolled onto this protocol).
  Young tumor infiltrating lymphocytes (TIL) + high dose aldesleukin
  Aldesleukin: Arm 1 - Days 1 to 4: Aldesleukin 720,000 IU/kg intravenous (IV) (based on total body weight) over 15 minutes every eight hours (+/- 1 hour) for up to 5 days (maximum 15 doses).
  Young TIL: Arm 1 - Day 0: Cells will be infused intravenously (IV) on the Patient Care Unit over 20-30 minutes.
Period: Overall Study
Arm/Group | Arm 1: Tumor Infiltrating Lymphocytes (TIL) + High Dose (HD) Interleukin-2 (IL-2) | Arm 2: Tumor Infiltrating Lymphocytes + High Dose Interleukin-2 + 1200 Total Body Irradiation (TBI) | Arm 1X: Tumor Infiltrating Lymphocytes (TIL) + High Dose (HD) Interleukin-2 (IL-2)
Started | 51 | 50 | 1
Completed | 51 | 48 | 1
Not Completed | 0 | 2 | 0
Not completed — Not treated: Rapid disease progression prior to start | 0 | 2 | 0

BASELINE CHARACTERISTICS:
Population: One participant on Arm 1X is not reported for privacy concerns (n=1).
Groups:
- Total: Total of all reporting groups
Arm/Group | Arm 1: Tumor Infiltrating Lymphocytes (TIL) + High Dose (HD) Interleukin-2 (IL-2) | Arm 2: Tumor Infiltrating Lymphocytes + High Dose Interleukin-2 + 1200 Total Body Irradiation (TBI) | Total
Number analyzed (Participants) | 51 | 50 | 101
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 50 | 50 | 100
  >=65 years | 1 | 0 | 1
Age, Continuous [Median (Inter-Quartile Range); unit: years] | 46.0 [36.9 to 54.2] | 47.1 [41.1 to 52.3] | 47.0 [39.2 to 54.1]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 17 | 20 | 37
  Male | 34 | 30 | 64
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Hispanic or Latino | 1 | 1 | 2
  Not Hispanic or Latino | 50 | 49 | 99
  Ethnicity Unknown or Not Reported | 0 | 0 | 0
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 1 | 1
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 0 | 2 | 2
  White | 50 | 46 | 96
  More than one race | 1 | 0 | 1
  Race Unknown or Not Reported | 1 | 1 | 2
Region of Enrollment [Number; unit: participants]
  United States | 51 | 50 | 101

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Participants Who Have a Clinical Response to Treatment (Objective Tumor Regression)
Description: Percentage of participants who have a clinical response to treatment (objective tumor regression) was measured by the Response Evaluation Criteria in Solid Tumors (RECIST) v1.0. Complete Response (CR) is disappearance of all target lesions. Partial Response (PR) is at least a 30% decrease in the sum of the longest diameter (LD) of target lesions taking as refence the baseline sum LD. Progressive Disease (PD) is at least a 20% increase in the sum of LD of target lesions taking as reference the smallest sum LD. The appearance of one or more new lesions is also considered progressions. Stable Disease (SD) is neither sufficient shrinkage to qualify for PR nor sufficient increase to qualify for PD taking as reference the smallest sum LD.
Time Frame: Participants were followed from treatment to progression of disease or until principal investigator (PI) discretion (average 91.8 months).
Population: 99/102 participants were analyzed. Two participants were not treated due to rapidly progressive disease after enrollment but before treatment. One participant on Arm 1X is not reported for privacy concerns (n=1).
Measure: Number; unit: Percentage of participants
Arm/Group | Arm 1: Tumor Infiltrating Lymphocytes (TIL) + High Dose (HD) Interleukin-2 (IL-2) | Arm 2: Tumor Infiltrating Lymphocytes + High Dose Interleukin-2 + 1200 Total Body Irradiation (TBI)
Number analyzed (Participants) | 51 | 48
Percentage of participants
  Complete Response | 27.5 | 27.1
  Partial Response | 19.6 | 37.5
  Stable Disease | 0 | 0
  Progressive Disease | 52.9 | 35.4

2. Primary Outcome: Overall Survival (OS)
Description: OS is defined as the time to death following the start of treatment.
Time Frame: Participants were followed from treatment until death (median 14 months) or until principal investigator (PI) discretion (median 99.0 months) for participants alive at study closure.
Population: 99/102 participants were analyzed. Two participants were enrolled and not treated due to rapid disease progression prior to start of treatment (Arm 2). One participant on Arm 1X is not reported for privacy concerns (n=1).
Measure: Median (Full Range); unit: Months
Groups:
- Arm 01: Tumor Infiltrating Lymphocytes (TIL) + High Dose (HD) Interleukin-2 (IL-2): Non-myeloablative lymphodepleting preparative regimen of cyclophosphamide and fludarabine + young tumor infiltrating lymphocytes (TIL) + high dose aldesleukin
  Aldesleukin: Arm 1 - Days 1 to 4: Aldesleukin 720,000 IU/kg intravenous (IV) (based on total body weight) over 15 minutes every eight hours (+/- 1 hour) for up to 5 days (maximum 15 doses).
  Cyclophosphamide: Arm 1 - Days -7 and -6: Cyclophosphamide 60 mg/kg/day X 2 days intravenous (IV) in 250 mL dextrose 5% in water (D5W) with Mesna 15 mg/kg/day X 2 days over 1 hr.
  Fludarabine: Arm 1 - Days -7 to -3: Fludarabine 25 mg/m^2/day intravenous piggyback (IVPB) daily over 15-30 minutes for 5 days.
  Young TIL: Arm 1 - Day 0: Cells will be infused intravenously (IV) on the Patient Care Unit over 20-30 minutes.
Arm/Group | Arm 01: Tumor Infiltrating Lymphocytes (TIL) + High Dose (HD) Interleukin-2 (IL-2) | Arm 2: Tumor Infiltrating Lymphocytes + High Dose Interleukin-2 + 1200 Total Body Irradiation (TBI)
Number analyzed (Participants) | 51 | 48
Months | 36.2 [1.2 to 158.3] | 37.3 [2.5 to 138.6]

3. Secondary Outcome: Progression-free Survival (PFS)
Description: PFS is defined as time to disease progression following the start of treatment. Disease progression was assessed by the Response Evaluation Criteria in Solid Tumors (RECIST) v3.0. Progressive Disease is at least a 20% increase in the sum of longest diameter (LD) of target lesions taking as reference the smallest sum LD. The appearance of one or more new lesions is also considered progression.
Time Frame: Participants were followed from treatment until death or until principal investigator (PI) discretion. A median of 91.8 months.
Population: as for outcome 2
Measure: Median (Full Range); unit: Months
Arm/Group | Arm 01: Tumor Infiltrating Lymphocytes (TIL) + High Dose (HD) Interleukin-2 (IL-2) | Arm 2: Tumor Infiltrating Lymphocytes + High Dose Interleukin-2 + 1200 Total Body Irradiation (TBI)
Number analyzed (Participants) | 51 | 48
Months | 6.8 [1.1 to 158.2] | 9.3 [0.5 to 109.9]

4. Secondary Outcome: Number of Grades 1, 2, 3, 4, and/or 5 Serious Adverse Events Possibly and/or Probably Related to Treatment
Description: Here is the number of Grades 2, 3, 4, and/or 5 serious adverse events possibly and/or probably related to treatment. Adverse events were assessed by the Common Terminology Criteria for Adverse Events (CTCAE v3.0). Grade 1 is mild. Grade 2 is moderate. Grade 3 is severe. Grade 4 is life-threatening. Grade 5 is death related to adverse event.
Time Frame: Time of registration through 6 years after the last treatment.
Population: 99/102 participants were analyzed. Two participants were enrolled and not treated due to disease progression prior to start of treatment (Arm 2). One participant on Arm 1X is not reported for privacy concerns (n=1). *Grade 1 and 2 adverse events were only captured when attributed to Young TIL or concurrently with other Grade ≥3 serious adverse events.
Measure: Number; unit: adverse events
Groups:
- Arm 1: Related to Interleukin-2 (IL-2); Arm 1: Related to Tumor Infiltrating Lymphocytes (TIL); Arm 1: Related to Fludarabine; Arm 1: Related to Cyclophosphamide: Arm 1: Tumor Infiltrating lymphocytes (TIL) + High Dose (HD) Interleukin-2 (IL-2) Non-myeloablative lymphodepleting preparative regimen of cyclophosphamide and fludarabine + young tumor infiltrating lymphocytes (TIL) + high dose aldesleukin
  Aldesleukin: Arm 1 - Days 1 to 4: Aldesleukin 720,000 IU/kg intravenous (IV) (based on total body weight) over 15 minutes every eight hours (+/- 1 hour) for up to 5 days (maximum 15 doses).
  Cyclophosphamide: Arm 1 - Days -7 and -6: Cyclophosphamide 60 mg/kg/day X 2 days intravenous (IV) in 250 mL dextrose 5% in water (D5W) with Mesna 15 mg/kg/day X 2 days over 1 hr.
  Fludarabine: Arm 1 - Days -7 to -3: Fludarabine 25 mg/m^2/day intravenous piggyback (IVPB) daily over 15-30 minutes for 5 days.
  Young TIL: Arm 1 - Day 0: Cells will be infused intravenously (IV) on the Patient Care Unit over 20-30 minutes.
- Arm 2: Related to Interleukin-2 (IL-2); Arm 2: Related to Tumor Infiltrating Lymphocytes; Arm 2: Related to Total Body Irradiation (TBI); Arm 2: Fludarabine; Arm 2: Related to Cyclophosphamide: Arm 2: Tumor Infiltrating lymphocytes + High Dose Interleukin-2 + 1200 Total Body Irradiation (TBI) Non-myeloablative lymphodepleting preparative regimen of cyclophosphamide and fludarabine + young tumor infiltrating lymphocytes (TIL) + high dose aldesleukin + total body irradiation (TBI)
  Aldesleukin: Arm 2 - Days 1 to 4: Aldesleukin 720,000 IU/kg intravenous (IV) (based on total body weight) over 15 minutes every eight hours (+/- 1 hour) for up to 5 days (maximum 15 doses).
  Cyclophosphamide: Arm 2 - Days -7 and -6: Cyclophosphamide 60 mg/kg/day X 2 days intravenous (IV) in 250 mL dextrose 5% in water (D5W) with Mesna 15 mg/kg/day X 2 days over 1 hr.
  Fludarabine: Arm 2 - Days -7 to -3: Fludarabine 25 mg/m^2/day intravenous piggyback (IVPB) daily over 15-30 minutes for 5 days.
  Young TIL: Arm 2 - Day 0: Cells will be infused intravenously (IV) on the Patient Care Unit over 20-30 minutes.
  Total Body Irradiation (TBI): Arm 2 - Days -3 to -1: Ondansetron 0.15 mg/kg intravenous (IV) x 1 dose pre-total body irradiation (TBI). Patients will then receive 2 Gray (Gy) TBI twice a day for 3 days (total dose 12 Gy using a linear accelerator in Radiation Oncology.
Arm/Group | Arm 1: Related to Interleukin-2 (IL-2) | Arm 1: Related to Tumor Infiltrating Lymphocytes (TIL) | Arm 1: Related to Fludarabine | Arm 1: Related to Cyclophosphamide | Arm 2: Related to Interleukin-2 (IL-2) | Arm 2: Related to Tumor Infiltrating Lymphocytes | Arm 2: Related to Total Body Irradiation (TBI) | Arm 2: Fludarabine | Arm 2: Related to Cyclophosphamide
Number analyzed (Participants) | 51 | 51 | 51 | 51 | 48 | 48 | 48 | 48 | 48
adverse events
  Any Grade 1 possibly and/or probably related | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Grade (Gr) 2 possibly related - Somnolence/depressed level of consciousness | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
  Grade 2 probably related - Supraventricular and nodal arrhythmia::Sinus tachycardia | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
  Grade 3 possibly related - Anorexia | 0 | 0 | 0 | 0 | 1 | 0 | 1 | 1 | 1
  Grade 3 probably related - Anorexia | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
  Grade 3 possibly related - Calcium, serum low (hypocalcemia) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
  Grade 3 possibly related - Creatinine | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1
  Grade 3 probably related - Creatinine | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
  Grade 3 probably related - Dyspnea (shortness of breath) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Grade 3 possibly related - left ventricular diastolic dysfunction | 0 | 0 | 0 | 0 | 1 | 0 | 1 | 1 | 1
  Grade 3 possibly related - Neurology - Other Specify, hydrocephalus | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
  Grade 3 possibly related - Pleural effusion (non-malignant) | 0 | 0 | 0 | 0 | 1 | 0 | 1 | 1 | 1
  Grade 3 possibly related - Renal failure | 1 | 0 | 0 | 0 | 1 | 1 | 0 | 1 | 1
  Grade 3 probably related - Renal failure | 0 | 0 | 1 | 1 | 0 | 0 | 0 | 0 | 0
  Grade 3 possibly related - Thrombotic microangiopathy (e.g., thrombotic thrombocytopenic purpura...) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
  Grade 3 probably related - Thrombotic microangiopathy (e.g., thrombotic thrombocytopenic purpura...) | 0 | 0 | 0 | 0 | 0 | 0 | 12 | 0 | 0
  Grade 4 probably related - Cardiopulmonary arrest, cause unknown (non-fatal) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
  Grade 4 possibly related - Infection (documented clinically or microbiologically) w/Grade 3 or 4 ANC | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Grade 4 probably related - Infection (documented clinically or microbiologically) w/Grade 3 or 4 ANC | 0 | 0 | 1 | 1 | 0 | 0 | 0 | 0 | 0
  Grade 4 probably related - Hemoglobin | 0 | 0 | 0 | 0 | 0 | 0 | 2 | 0 | 0
  Grade 4 possibly related - Hemolysis (e.g., immune hemolytic anemia, drug-related hemolysis) | 0 | 0 | 0 | 0 | 1 | 0 | 1 | 1 | 1
  Grade 4 possibly related - Secondary Malignancy - possibly related to cancer treatment (Specify, __) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 1
  Any Grade 5 possibly and/or probably related | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0

5. Secondary Outcome: Number of Grades 1, 2, 3, 4, and/or 5 Non-serious Adverse Events Possibly and/or Probably Related to Treatment
Description: Here is the number of Grades 1, 2, 3, 4, and/or 5 non-serious adverse events possibly and/or probably related to treatment. Adverse events were assessed by the Common Terminology Criteria for Adverse Events (CTCAE v3.0). Grade 1 is mild. Grade 2 is moderate. Grade 3 is severe. Grade 4 is life-threatening. Grade 5 is death related to adverse event.
Time Frame: 30 days after end of treatment, up to 6 years
Population: as for outcome 4
Measure: Number; unit: adverse events
Arm/Group | Arm 1: Related to Interleukin-2 (IL-2) | Arm 1: Related to Tumor Infiltrating Lymphocytes (TIL) | Arm 1: Related to Fludarabine | Arm 1: Related to Cyclophosphamide | Arm 2: Related to Interleukin-2 (IL-2) | Arm 2: Related to Tumor Infiltrating Lymphocytes | Arm 2: Related to Total Body Irradiation (TBI) | Arm 2: Fludarabine | Arm 2: Related to Cyclophosphamide
Number analyzed (Participants) | 51 | 51 | 51 | 51 | 48 | 48 | 48 | 48 | 48
adverse events
  Grade 1 probably related - Confusion | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
  Grade 1 possibly related - Diarrhea | 0 | 0 | 0 | 0 | 1 | 0 | 1 | 1 | 1
  Grade 1 probably related - Mood alteration::Agitation | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
  Grade 1 probably related - Dyspnea (shortness of breath) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Grade 1 Fatigue (asthenia, lethargy, malaise) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Grade 1 possibly related - Hypopigmentation | 2 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Grade 1 probably related - Hypopigmentation | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Grade 1 Pain::Chest wall | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
  Grade 1 probably related - Renal/Genitourinary - Other (Specify, Lower urine output) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Grade 2 probably related - Acute vascular leak syndrome | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Grade 2 probably related - Confusion | 4 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
  Grade 2 possibly related - Creatinine | 0 | 0 | 1 | 1 | 1 | 0 | 0 | 1 | 1
  Grade 2 probably related - Creatinine | 1 | 0 | 0 | 0 | 3 | 0 | 0 | 0 | 0
  Grade 2 probably related - Diarrhea | 1 | 0 | 1 | 1 | 2 | 0 | 1 | 1 | 1
  Grade 2 possibly related - Dry mouth/salivary gland (xerostomia) | 0 | 0 | 0 | 0 | 1 | 0 | 1 | 0 | 0
  Grade 2 possibly related - Dyspnea (shortness of breath) | 1 | 1 | 1 | 1 | 0 | 1 | 0 | 0 | 0
  Grade 2 probably related - Dyspnea (shortness of breath) | 13 | 0 | 0 | 0 | 12 | 1 | 0 | 0 | 0
  Grade 2 possibly related - Fatigue | 1 | 0 | 10 | 10 | 1 | 0 | 6 | 6 | 6
  Grade 2 probably related - Hemorrhage, GU:: Bladder | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
  Grade 2 - possibly related - hypopigmentation | 0 | 1 | 0 | 0 | 1 | 1 | 0 | 0 | 0
  Grade 2 - probably related - hypopigmentation | 4 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
  Grade 2 probably related - Hypotension | 7 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Grade 2 possibly related - Hypoxia | 0 | 0 | 0 | 0 | 4 | 1 | 0 | 0 | 0
  Grade 2 probably related - Mental status | 1 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
  Grade 2 probably related - Mood alteration::Agitation | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
  Grade 2 probably related - Neuropathy:sensory | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
  Grade 2 possibly related - Ocular/Visual - Other, Specify (Corneal Edema, OU) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
  Grade 2 probably related - Psychosis (hallucinations/delusions) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
  Grade 2 probably related - Rash/desquamation | 2 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Grade 2 probably related - Renal/Genitourinary - Other (Specify, Lower urine output) | 2 | 0 | 0 | 0 | 3 | 0 | 0 | 0 | 0
  Grade 2 possibly related - Rigors/chills | 0 | 0 | 0 | 0 | 1 | 1 | 0 | 0 | 0
  Grade 2 probably related - Somnolence/depressed level of consciousness | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
  Grade 2 possibly related - Supraventricular and nodal arrhythmia::Atrial fibrillation | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1
  Grade 2 possibly related - Uveitis | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Grade 2 possibly related - Vision-blurred vision | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
  Grade 3 possibly related - Acidosis (metabolic or respiratory) | 0 | 0 | 0 | 0 | 1 | 0 | 1 | 1 | 1
  Grade 3 possibly related - Acute vascular leak syndrome | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1
  Grade 3 probably related - Acute vascular leak syndrome | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Grade 3 possibly related - Albumin, serum-low (hypoalbuminemia) | 1 | 0 | 2 | 2 | 0 | 0 | 0 | 2 | 2
  Grade 3 probably related - Albumin, serum-low (hypoalbuminemia) | 1 | 0 | 2 | 2 | 2 | 0 | 0 | 0 | 0
  Grade 3 possibly related - Alkaline phosphatase | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 1 | 1
  Grade 3 possibly related - ALT, SGPT (serum glutamic pyruvic transaminase) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 2 | 2
  Grade 3 probably related - ALT, SGPT (serum glutamic pyruvic transaminase) | 0 | 0 | 1 | 1 | 0 | 0 | 0 | 2 | 2
  Grade 3 possibly related - Anorexia | 0 | 0 | 0 | 0 | 1 | 0 | 1 | 1 | 1
  Grade 3 possibly related - AST, SGOT(serum glutamic oxaloacetic transaminase) | 1 | 0 | 1 | 1 | 1 | 0 | 0 | 1 | 1
  Grade 3 probably related - AST, SGOT(serum glutamic oxaloacetic transaminase) | 1 | 0 | 2 | 2 | 0 | 0 | 0 | 1 | 1
  Grade 3 possibly related - Bilirubin (hyperbilirubinemia) | 1 | 0 | 2 | 2 | 1 | 0 | 1 | 1 | 1
  Grade 3 possibly related - Calcium, serum low (hypocalcemia) | 0 | 0 | 0 | 0 | 1 | 0 | 1 | 2 | 2
  Grade 3 probably related - Calcium, serum low (hypocalcemia) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 2 | 2
  Grade 3 probably related - Cardiac troponin I (cTnl) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
  Grade 3 probably related - Colitis, infectious (e.g., Clostridium difficile) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1
  Grade 3 probably related - Creatinine | 1 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
  Grade 3 probably related - Diarrhea | 0 | 0 | 0 | 0 | 1 | 0 | 3 | 3 | 3
  Grade 3 possibly related - Dry mouth/salivary gland (xerostomia) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 1
  Grade 3 probably related - Dry mouth/salivary gland (xerostomia) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
  Grade 3 possibly related - Dyspnea (shortness of breath) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
  Grade 3 probably related - Dyspnea (shortness of breath) | 9 | 0 | 1 | 1 | 5 | 0 | 0 | 0 | 0
  Grade 3 possibly related - Edema: head and neck | 1 | 0 | 1 | 1 | 0 | 0 | 0 | 0 | 0
  Grade 3 possibly related - Fatigue (asthenia, lethargy, malaise) | 0 | 0 | 2 | 2 | 2 | 0 | 5 | 2 | 2
  Grade 3 probably related - Fatigue (asthenia, lethargy, malaise) | 2 | 0 | 0 | 0 | 4 | 0 | 1 | 4 | 4
  Grade 3 possibly related - Febrile neutropenia | 1 | 0 | 0 | 0 | 1 | 0 | 4 | 0 | 0
  Grade 3 probably related - Febrile neutropenia | 0 | 0 | 23 | 23 | 0 | 0 | 0 | 35 | 35
  Grade 3 possibly related - Fever | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1
  Grade 3 probably related - Fever | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1
  Grade 3 possibly related - Hemoglobin | 12 | 0 | 9 | 9 | 13 | 0 | 12 | 16 | 16
  Grade 3 probably related - Hemoglobin | 0 | 0 | 13 | 13 | 2 | 0 | 0 | 18 | 18
  Grade 3 possibly related - Hemorrhage, GI::Ileum | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
  Grade 3 probably related - Hemorrhage, GI::Ileum | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1
  Grade 3 probably related - Hypotension | 2 | 0 | 0 | 0 | 3 | 0 | 0 | 0 | 0
  Grade 3 possibly related - Hypoxia | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Grade 3 probably related - Hypoxia | 10 | 1 | 1 | 1 | 10 | 0 | 0 | 0 | 0
  Grade 3 possibly related - Infection (documented clinically or microbiologically)..Blood | 1 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
  Grade 3 probably related - Infection (documented clinically or microbiologically)...Blood | 0 | 0 | 1 | 1 | 0 | 0 | 0 | 2 | 2
  Grade 3 possibly related - Infection with normal ANC or Grade 1 or 2 neutrophils::Blood | 1 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
  Grade 3 probably related - Infection with normal ANC or Grade 1 or 2 neutrophils::Blood | 0 | 0 | 1 | 1 | 1 | 0 | 0 | 2 | 2
  Grade 3 probably related- Infection (documented clinically or microbiologically)...Urinary tract NOS | 0 | 0 | 1 | 1 | 0 | 0 | 0 | 2 | 2
  Grade 3 probably related - Infection with normal ANC or Grade 1 or 2 neutrophils::Upper airway NOS | 0 | 0 | 1 | 1 | 1 | 0 | 0 | 0 | 0
  Grade 3 probably related - Infection with normal ANC or Grade 1 or 2 neutrophils::Urinary tract NOS | 0 | 0 | 1 | 1 | 0 | 0 | 0 | 2 | 2
  Grade 3 possibly related - Infection with normal ANC or Grade 1 or 2 neutrophils::Skin (cellulitis) | 0 | 0 | 1 | 1 | 0 | 0 | 0 | 0 | 0
  Grade 3 possibly related - Leukocytes (total WBC) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1
  Grade 3 probably related - Leukocytes (total WBC) | 0 | 0 | 1 | 1 | 0 | 0 | 0 | 0 | 0
  Grade 3 possibly related - Lymphopenia | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1
  Grade 3 probably related - Lymphopenia | 0 | 0 | 2 | 2 | 0 | 0 | 0 | 0 | 0
  Grade 3 possibly related - Mental status | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
  Grade 3 possibly related - Mucositis/stomatitis (clinical exam)::Oral cavity | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1
  Grade 3 probably related - Mucositis/stomatitis (clinical exam)::Oral cavity | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 1
  Grade 3 possibly related - Nausea | 1 | 0 | 0 | 0 | 3 | 0 | 3 | 2 | 2
  Grade 3 probably related - Nausea | 0 | 0 | 2 | 2 | 3 | 0 | 4 | 9 | 9
  Grade 3 possibly related - Neutrophils/granulocytes (ANC/AGC) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
  Grade 3 probably related - Neutrophils/granulocytes (ANC/AGC) | 0 | 0 | 1 | 1 | 0 | 0 | 0 | 4 | 4
  Grade 3 possibly related - Pain::Abdomen NOS | 0 | 0 | 2 | 2 | 1 | 0 | 0 | 1 | 1
  Grade 3 probably related - Pain::Abdomen NOS | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
  Grade 3 probably related - Pain::Bladder | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
  Grade 3 possibly related - Pain::Chest/thorax NOS | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
  Grade 3 possibly related - Pain::Head/headache | 3 | 0 | 7 | 7 | 1 | 0 | 0 | 2 | 2
  Grade 3 possibly related - Pain::Joint | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1
  Grade 3 possibly related - Pain::Muscle | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
  Grade 3 possibly related - Pain::Pain NOS | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 3 | 3
  Grade 3 possibly related - Phosphate, serum-low (hypophosphatemia) | 4 | 0 | 10 | 10 | 11 | 0 | 2 | 12 | 12
  Grade 3 probably related - Phosphate, serum-low (hypophosphatemia) | 1 | 0 | 3 | 3 | 2 | 0 | 0 | 2 | 3
  Grade 3 probably related - Platelets | 0 | 0 | 4 | 4 | 0 | 0 | 0 | 1 | 1
  Grade 3 possibly related - Pleural effusion | 1 | 0 | 1 | 1 | 1 | 0 | 0 | 1 | 1
  Grade 3 possibly related - Pneumonitis/pulmonary infiltrates | 0 | 0 | 1 | 1 | 0 | 0 | 0 | 0 | 0
  Grade 3 probably related - Pneumonitis/pulmonary infiltrates | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
  Grade 3 possibly related - Potassium, serum-low (hypokalemia) | 0 | 0 | 0 | 0 | 2 | 0 | 2 | 2 | 2
  Grade 3 probably related - Potassium, serum-low (hypokalemia) | 0 | 0 | 0 | 0 | 2 | 0 | 0 | 1 | 1
  Grade 3 probably related - Psychosis | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
  Grade 3 possibly related - PTT (Partial Thromboplastin Time) | 1 | 0 | 1 | 1 | 0 | 0 | 0 | 2 | 2
  Grade 3 probably related - PTT (Partial Thromboplastin Time) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
  Grade 3 possibly related - Rash/desquamation | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Grade 3 probably related - Rash/desquamation | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
  Grade 3 possibly related - Renal failure | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
  Grade 3 probably related - Renal/Genitourinary - Other (Specify, Oliguria) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Grade 3 probably related - Renal failure | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
  Grade 3 possibly related - Retinopathy | 0 | 0 | 1 | 1 | 0 | 0 | 0 | 0 | 0
  Grade 3 possibly related - Rigors/chills | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1
  Grade 3 probably related - Rigors/chills | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
  Grade 3 possibly related - Sodium, serum-low (hyponatremia) | 1 | 0 | 1 | 1 | 2 | 0 | 1 | 1 | 1
  Grade 3 possibly related - Supraventricular and nodal arrhythmia::Atrial fibrillation | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1
  Grade 3 probably related - Supraventricular and nodal arrhythmia::Atrial fibrillation | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
  Grade 3 possibly related - Supraventricular and nodal arrhythmia::Sinus bradycardia | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
  Grade 3 probably related - Supraventricular and nodal arrhythmia::Sinus tachycardia | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
  Grade 3 possibly related - Syncope (fainting) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 1 | 1
  Grade 3 probably related - Syncope (fainting) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
  Grade 3 probably related - Thrombotic microangiopathy | 0 | 0 | 0 | 0 | 0 | 0 | 5 | 0 | 0
  Grade 3 possibly related - Vomiting | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
  Grade 3 probably related - Vomiting | 0 | 0 | 0 | 0 | 2 | 0 | 0 | 2 | 2
  Grade 4 probably related - Bilirubin (hyperbilirubinemia) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1
  Grade 4 possibly related - Calcium, serum-low (hypocalcemia) | 0 | 0 | 0 | 0 | 1 | 0 | 1 | 1 | 1
  Grade 4 probably related - Calcium, serum-low (hypocalcemia) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1
  Grade 4 probably related - Febrile neutropenia | 0 | 0 | 2 | 2 | 0 | 0 | 0 | 3 | 3
  Grade 4 possibly related - Hypotension | 0 | 0 | 0 | 0 | 1 | 0 | 1 | 1 | 1
  Grade 4 possibly related - Infection with normal ANC or Grade 1 or 2 neutrophils::Blood | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1
  Grade 4 probably related - Infection with normal ANC or Grade 1 or 2 neutrophils::Blood | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
  Grade 4 possibly related - Infection with normal ANC or Grade 1 or 2 neutrophils::Trachea | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1
  Grade 4 probably related - Infection with normal ANC or Grade 1 or 2 neutrophils::Trachea | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
  Grade 4 possibly related - Infection with normal ANC or Grade 1 or 2 neutrophils Urinary tract NOS | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1
  Grade 4 probably related - Infection with normal ANC or Grade 1 or 2 neutrophils::Urinary tract NOS | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
  Grade 4 possibly related - Leukocytes (total WBC) | 1 | 0 | 0 | 0 | 1 | 0 | 13 | 0 | 0
  Grade 4 probably related - Leukocytes (total WBC) | 0 | 0 | 50 | 50 | 0 | 0 | 0 | 48 | 48
  Grade 4 possibly related - Lymphopenia | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
  Grade 4 probably related - Lymphopenia | 0 | 0 | 51 | 51 | 0 | 0 | 0 | 48 | 48
  Grade 4 possibly related - Neutrophils/granulocytes (ANC/AGC) | 1 | 0 | 1 | 1 | 1 | 0 | 11 | 0 | 0
  Grade 4 probably related - Neutrophils/granulocytes (ANC/AGC) | 0 | 0 | 50 | 50 | 0 | 0 | 0 | 46 | 46
  Grade 4 probably related - Phosphate, serum-low (hypophosphatemia) | 0 | 0 | 1 | 1 | 0 | 0 | 0 | 0 | 0
  Grade 4 possibly related - Platelets | 1 | 0 | 0 | 0 | 1 | 0 | 15 | 0 | 0
  Grade 4 probably related - Platelets | 0 | 0 | 39 | 39 | 0 | 0 | 0 | 39 | 39
  Grade 4 possibly related - Potassium, serum-low (hypokalemia) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 1 | 1
  Grade 4 probably relatedRenal/Genitourinary-Other (Low urine output(nonoliguric renal insufficiency) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0

6. Other Pre Specified Outcome: Number of Participants With Serious and/or Non-serious Adverse Events Assessed by the Common Terminology Criteria for Adverse Events (CTCAE v3.0)
Description: Here is the number of participants with serious and/or non-serious adverse events assessed by the Common Terminology Criteria for Adverse Events (CTCAE v3.0). A non-serious adverse event is any untoward medical occurrence. A serious adverse event is an adverse event or suspected adverse reaction that results in death, a life-threatening adverse drug experience, hospitalization, disruption of the ability to conduct normal life functions, congenital anomaly/birth defect or important medical events that jeopardize the patient or subject and may require medical or surgical intervention to prevent one of the previous outcomes mentioned.
Time Frame: Participants will be followed for adverse events from registration through 30 days after the last treatment, up to 6 years
Population: as for outcome 4
Measure: Count of Participants; unit: Participants
Arm/Group | Arm 01: Tumor Infiltrating Lymphocytes (TIL) + High Dose (HD) Interleukin-2 (IL-2) | Arm 2: Tumor Infiltrating Lymphocytes + High Dose Interleukin-2 + 1200 Total Body Irradiation (TBI)
Number analyzed (Participants) | 51 | 48
Participants | 51 | 48

ADVERSE EVENTS:
Time Frame: All-Cause Mortality was monitored/assessed from treatment to study closure (median 12.3 years). Adverse events were monitored/assessed from start of treatment until 30 days after the last treatment, up to 6 years.
Description: 99/102 participants were analyzed for Adverse Events. Two participants were enrolled/not treated (Arm 2). One participant on Arm 1X is not reported for privacy concerns (n=1). *Grade 1 and 2 adverse events were only captured when attributed to Young TIL or concurrently with other Grade ≥3 serious adverse events.
Arm/Group | Arm 1: Tumor Infiltrating Lymphocytes (TIL) + High Dose (HD) Interleukin-2 (IL-2) | Arm 2: Tumor Infiltrating Lymphocytes + High Dose Interleukin-2 + 1200 Total Body Irradiation (TBI)
All-Cause Mortality (participants affected / at risk) | 23/51 | 23/50
Serious Adverse Events (participants affected / at risk) | 2/51 | 17/48
Other Adverse Events (participants affected / at risk) | 51/51 | 48/48
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Arm 1: Tumor Infiltrating Lymphocytes (TIL) + High Dose (HD) Interleukin-2 (IL-2) (N=51) | Arm 2: Tumor Infiltrating Lymphocytes + High Dose Interleukin-2 + 1200 Total Body Irradiation (TBI) (N=48)
Allergic reaction/hypersensitivity (including drug fever) (Immune system disorders) | 0 (0) | 1 (1)
Anorexia (Gastrointestinal disorders) | 0 (0) | 2 (2)
Calcium, serum-low (hypocalcemia) (Metabolism and nutrition disorders) | 0 (0) | 1 (1)
Cardiopulmonary arrest, cause unknown (non-fatal) (Cardiac disorders) | 0 (0) | 1 (1)
Creatinine (Metabolism and nutrition disorders) | 0 (0) | 1 (1)
Death not associated with CTCAE term (General disorders) | 0 (0) | 1 (1)
Death not associated with CTCAE term::Disease progression NOS (General disorders) | 1 (1) | 0 (0)
Dyspnea (shortness of breath) (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Hemoglobin (Blood and lymphatic system disorders) | 0 (0) | 2 (2)
Hemolysis (e.g., immune hemolytic anemia, drug-related hemolysis) (Blood and lymphatic system disorders) | 0 (0) | 1 (1)
Infection (Infections and infestations) | 1 (1) | 0 (0) — (documented clinically or microbiologically) with Grade 3 or 4 neutrophils (ANC <1.0 x 10e9/L)::Blood
Left ventricular diastolic dysfunction (Cardiac disorders) | 0 (0) | 1 (1)
Neurology - Other (Specify, __): HYDROCEPHALUS (Nervous system disorders) | 0 (0) | 1 (1)
Pleural effusion (non-malignant) (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Renal failure (Renal and urinary disorders) | 1 (1) | 1 (1)
Secondary Malignancy (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1) — - possibly related to cancer treatment (Specify, __): Myelodysplastic syndrome versus acute myeloid leukemia
Seizure (Nervous system disorders) | 0 (0) | 1 (1)
Somnolence/depressed level of consciousness (Nervous system disorders) | 0 (0) | 1 (1)
Supraventricular and nodal arrhythmia::Sinus tachycardia (Cardiac disorders) | 0 (0) | 1 (1)
Syncope (fainting) (Nervous system disorders) | 0 (0) | 1 (1)
Thrombosis/embolism (vascular access-related) (Vascular disorders) | 0 (0) | 1 (1)
Thrombosis/thrombus/embolism (Vascular disorders) | 0 (0) | 1 (1)
Thrombotic microangiopathy (Blood and lymphatic system disorders) | 0 (0) | 8 (8) — (e.g., thrombotic thrombocytopenic purpura [TTP] or hemolytic uremic syndrome [HUS])
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Arm 1: Tumor Infiltrating Lymphocytes (TIL) + High Dose (HD) Interleukin-2 (IL-2) (N=51) | Arm 2: Tumor Infiltrating Lymphocytes + High Dose Interleukin-2 + 1200 Total Body Irradiation (TBI) (N=48)
ALT, SGPT (serum glutamic pyruvic transaminase) (Metabolism and nutrition disorders) | 1 (1) | 4 (4)
AST, SGOT(serum glutamic oxaloacetic transaminase) (Metabolism and nutrition disorders) | 4 (4) | 3 (4)
Acidosis (metabolic or respiratory) (Metabolism and nutrition disorders) | 0 (0) | 1 (1)
Acute vascular leak syndrome (Vascular disorders) | 3 (3) | 2 (2)
Adrenal insufficiency (Endocrine disorders) | 0 (0) | 1 (1)
Albumin, serum-low (hypoalbuminemia) (Metabolism and nutrition disorders) | 4 (6) | 12 (12)
Alkaline phosphatase (Metabolism and nutrition disorders) | 0 (0) | 2 (2)
Anorexia (Gastrointestinal disorders) | 0 (0) | 1 (1)
Bilirubin (hyperbilirubinemia) (Metabolism and nutrition disorders) | 2 (2) | 2 (2)
Calcium, serum-low (hypocalcemia) (Metabolism and nutrition disorders) | 0 (0) | 7 (8)
Cardiac troponin I (cTnI) (Cardiac disorders) | 0 (0) | 1 (1)
Colitis, infectious (e.g., Clostridium difficile) (Infections and infestations) | 0 (0) | 1 (1)
Confusion (Nervous system disorders) | 3 (3) | 2 (2)
Creatinine (Metabolism and nutrition disorders) | 4 (4) | 5 (5)
Diarrhea (Gastrointestinal disorders) | 1 (1) | 5 (5)
Dry mouth/salivary gland (xerostomia) (Gastrointestinal disorders) | 0 (0) | 2 (2)
Dyspnea (shortness of breath) (Respiratory, thoracic and mediastinal disorders) | 24 (24) | 18 (20)
Edema: head and neck (Blood and lymphatic system disorders) | 1 (1) | 0 (0)
Fatigue (asthenia, lethargy, malaise) (General disorders) | 17 (17) | 14 (14)
Febrile neutropenia (Infections and infestations) | 26 (26) | 36 (38) — (fever of unknown origin without clinically or microbiologically documented infection)(ANC <1.0 x 10e9/L, fever >=38.5 degrees C)
Fever (in the absence of neutropenia, where neutropenia is defined as ANC <1.0 x 10e9/L) (General disorders) | 0 (0) | 3 (3)
Hemoglobin (Blood and lymphatic system disorders) | 20 (22) | 31 (35)
Hemorrhage, GI::Ileum (Gastrointestinal disorders) | 0 (0) | 1 (1)
Hemorrhage, GU::Bladder (Renal and urinary disorders) | 1 (1) | 0 (0)
Hypopigmentation (Skin and subcutaneous tissue disorders) | 8 (8) | 2 (2)
Hypotension (Cardiac disorders) | 10 (10) | 9 (9)
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 12 (12) | 11 (12)
Incontinence, urinary (Renal and urinary disorders) | 1 (1) | 0 (0)
Infection (Infections and infestations) | 12 (13) | 5 (6) — (documented clinically or microbiologically) with Grade 3 or 4 neutrophils (ANC <1.0 x 10e9/L)::Blood
Infection (Infections and infestations) | 0 (0) | 2 (2) — (documented clinically or microbiologically) with Grade 3 or 4 neutrophils (ANC <1.0 x 10e9/L)::Urinary tract NOS
Infection with normal ANC or Grade 1 or 2 neutrophils::Blood (Infections and infestations) | 1 (1) | 3 (3)
Infection with normal ANC or Grade 1 or 2 neutrophils::Skin (cellulitis) (Infections and infestations) | 0 (0) | 1 (1)
Infection with normal ANC or Grade 1 or 2 neutrophils::Trachea (Infections and infestations) | 0 (0) | 1 (1)
Infection with normal ANC or Grade 1 or 2 neutrophils::Upper airway NOS (Infections and infestations) | 1 (1) | 0 (0)
Infection with normal ANC or Grade 1 or 2 neutrophils::Urinary tract NOS (Infections and infestations) | 1 (1) | 3 (3)
Infection with unknown ANC::Nerve-peripheral (Infections and infestations) | 0 (0) | 1 (1)
Leukocytes (total WBC) (Blood and lymphatic system disorders) | 51 (51) | 48 (49)
Lymphopenia (Blood and lymphatic system disorders) | 51 (55) | 48 (50)
Mental status (Nervous system disorders) | 2 (2) | 2 (2)
Mood alteration::Agitation (Nervous system disorders) | 0 (0) | 2 (2)
Mucositis/stomatitis (clinical exam)::Oral cavity (Gastrointestinal disorders) | 0 (0) | 1 (1)
Muscle weakness, generalized or specific area (not due to neuropathy)::Extremity-upper (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Nausea (Gastrointestinal disorders) | 2 (2) | 9 (9)
Neuropathy: sensory (Nervous system disorders) | 1 (1) | 0 (0)
Neutrophils/granulocytes (ANC/AGC) (Blood and lymphatic system disorders) | 51 (51) | 48 (48)
Ocular/Visual - Other (Specify, __): Corneal Edema, OU (Eye disorders) | 0 (0) | 1 (1)
Ocular/Visual - Other (Specify, __): VISION CHANGES (R EYE) (Eye disorders) | 1 (1) | 0 (0)
PTT (Partial Thromboplastin Time) (Blood and lymphatic system disorders) | 1 (1) | 3 (4)
Pain::Abdomen NOS (Gastrointestinal disorders) | 2 (2) | 1 (1)
Pain::Back (Musculoskeletal and connective tissue disorders) | 0 (0) | 2 (2)
Pain::Bladder (Renal and urinary disorders) | 1 (1) | 0 (0)
Pain::Breast (Reproductive system and breast disorders) | 1 (1) | 0 (0)
Pain::Chest wall (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 1 (1)
Pain::Chest/thorax NOS (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Pain::Extremity-limb (Musculoskeletal and connective tissue disorders) | 2 (2) | 0 (0)
Pain::Face (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
Pain::Head/headache (Nervous system disorders) | 7 (7) | 2 (2)
Pain::Joint (Musculoskeletal and connective tissue disorders) | 0 (0) | 2 (2)
Pain::Muscle (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Pain::Neuralgia/peripheral nerve (Nervous system disorders) | 0 (0) | 1 (2)
Pain::Pain NOS (General disorders) | 0 (0) | 2 (2)
Pain::Pelvis (Reproductive system and breast disorders) | 1 (1) | 0 (0)
Pain::Sinus (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Pain::Tumor pain (General disorders) | 1 (1) | 0 (0)
Phosphate, serum-low (hypophosphatemia) (Metabolism and nutrition disorders) | 13 (15) | 15 (18)
Platelets (Blood and lymphatic system disorders) | 40 (40) | 39 (40)
Pleural effusion (non-malignant) (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 1 (1)
Pneumonitis/pulmonary infiltrates (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 1 (1)
Potassium, serum-low (hypokalemia) (Metabolism and nutrition disorders) | 0 (0) | 5 (5)
Pruritus/itching (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
Psychosis (hallucinations/delusions) (Nervous system disorders) | 5 (5) | 7 (7)
Rash/desquamation (Skin and subcutaneous tissue disorders) | 5 (5) | 2 (2)
Renal failure (Renal and urinary disorders) | 0 (0) | 2 (2)
Renal/Genitourinary - Other (Specify, __): Low urine output (Renal and urinary disorders) | 0 (0) | 3 (3)
Renal/Genitourinary - Other (Specify, __): Low urine output (nonoliguric renal insufficiency) (Renal and urinary disorders) | 1 (1) | 0 (0)
Renal/Genitourinary - Other (Specify, __): Lower urine output (Renal and urinary disorders) | 3 (3) | 0 (0)
Renal/Genitourinary - Other (Specify, __): Oliguria (Renal and urinary disorders) | 1 (1) | 0 (0)
Renal/Genitourinary - Other (Specify, __): low urine output (Renal and urinary disorders) | 0 (0) | 1 (1)
Retinopathy (Eye disorders) | 1 (1) | 0 (0)
Rigors/chills (General disorders) | 0 (0) | 2 (2)
Sodium, serum-low (hyponatremia) (Metabolism and nutrition disorders) | 1 (1) | 3 (3)
Somnolence/depressed level of consciousness (Nervous system disorders) | 0 (0) | 1 (1)
Supraventricular and nodal arrhythmia::Atrial fibrillation (Cardiac disorders) | 2 (2) | 4 (4)
Supraventricular and nodal arrhythmia::Sinus bradycardia (Cardiac disorders) | 0 (0) | 1 (1)
Supraventricular and nodal arrhythmia::Sinus tachycardia (Cardiac disorders) | 0 (0) | 1 (1)
Syncope (fainting) (Nervous system disorders) | 0 (0) | 3 (3)
Thrombotic microangiopathy (Blood and lymphatic system disorders) | 0 (0) | 5 (5) — (e.g., thrombotic thrombocytopenic purpura [TTP] or hemolytic uremic syndrome [HUS])
Urinary frequency/urgency (Renal and urinary disorders) | 0 (0) | 1 (1)
Uveitis (Eye disorders) | 1 (1) | 0 (0)
Ventricular arrhythmia::Ventricular tachycardia (Cardiac disorders) | 0 (0) | 1 (1)
Vision-blurred vision (Eye disorders) | 0 (0) | 1 (1)
Vision-flashing lights/floaters (Eye disorders) | 1 (1) | 0 (0)
Vomiting (Gastrointestinal disorders) | 0 (0) | 2 (2)

LIMITATIONS AND CAVEATS:
Grade 1/2 adverse events were only captured in conjunction with serious adverse events or when attributed to TIL.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2022-04-15): https://cdn.clinicaltrials.gov/large-docs/65/NCT01319565/Prot_SAP_000.pdf
  • Informed Consent Form (2019-04-09): https://cdn.clinicaltrials.gov/large-docs/65/NCT01319565/ICF_001.pdf